CLINICAL TRIAL: NCT02078414
Title: Continued Use of Effective Contraception After Use of Emergency Contraception
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Helena Kopp Kallner, Consultant Obstetrics and Gynecology, PhD, Karolinska Institutet
Other Study IDs: RFSU1
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Emergency Contraception; Contraception; Reproductive Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Ulipristal acetate: Women choosing EllaOne as emergency contraception
- Copper IUD: Women choosing copper IUD as emergency contraception

SUMMARY:
Women using an emergency contraceptive method must use back up protection for 1-2 weeks depending on method. The Copper-IUD is the most effective emergency contraceptive method. The investigators wish to explore if women choosing the Cooper IUD have a higher frequency of use of an effective contraceptive method 3 months and 6 months after the use of an emergency contraceptive method than women who choose to use the emergency contraceptive pill EllaOne (ulipristal acetate).

ELIGIBILITY:
Inclusion Criteria:

* women over 18 years
* eligible for all emergency contraception

Exclusion Criteria:

* previous conisation
* known stenosis of the cervix
* signs of ongoing genital infection
* known uterine anomaly
* Known bleeding disorder

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women without contraception or with a failed contraceptive method seeking emergency contraception
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2014-03; Primary Completion 2015-02 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Use of an effective contraceptive method | 6 months after emergency contraceptive use
  Use of pill, patch, ring, IUD, IUS, or injection 6 months after use of emergency contraceptive method

CONTACTS AND LOCATIONS:
Locations (1):
- RFSU clinic, Stockholm, Sweden